CLINICAL TRIAL: NCT06965491
Title: Exploring the Role of Intermittent Exogenous Ketosis on Physical and Mental Fatigue During Ultra-endurance Performance
Brief Title: The Effects of Exogenous Ketosis on Ultra-endurance Recovery and Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Chiel Poffé, Assistant Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: S68178
Record Dates: First submitted 2024-10-04; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Exogenous Ketosis; Endurance Cycling Performance; Fatigue; Muscle, Heart; Fatigue, Mental
Keywords: ultra-endurance; cycling; physiological strain; mental fatigue
MeSH Terms: conditions — Fatigue; Mental Fatigue

STUDY DESIGN:
Intervention Model Description: Riders will be paired matched and randomly assigned to either the ketone ester supplementation (KE) group or the control group (CON) which will receive an isocaloric taste-matched placebo
Who Masked: Participant, Investigator
Masking Description: Participants and investigators are blinded from the experimental condition (KE or CON). Supplements are provided in non transparent tubes and the control supplement is identical in taste and viscosity to the ketone supplement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): Intervention: 8-day multistage mountain bike race/simulation Dietary intervention: placebo supplement (oral supplement containing: 16.4 grams of medium chained triglycerides, 1mM of sucrose octaacetate and water)
  Interventions: Dietary Supplement: Placebo Supplement
- Experimental group (Experimental): Intervention: 8-day multistage mountain bike race/simulation Dietary intervention: ketone ester supplement (25 grams of pure R-(3)-hydroxybutyl-(R)-3-hydroxybutyrate ketone monoester drink)
  Interventions: Dietary Supplement: Ketone ester supplement

INTERVENTIONS:
Dietary Supplement: Placebo Supplement — Placebo supplement:
  Oral supplement containing: 16.4 grams of medium chained triglycerides, 1mM or sucrose octaacetate and water
  Arms: Control group
Dietary Supplement: Ketone ester supplement — Ketone ester supplement Oral supplement containing: 25 grams of pure (R)-3-hydroxybutyl-(R)-3-hydroxybutyrate ketone monoester drink
  Arms: Experimental group

SUMMARY:
The study aims to investigate the effects of post-exercise and pre-sleep ketosis via oral ketone ester supplementation on physical and mental recovery during a multi-day cycling stage race.

DETAILED DESCRIPTION:
Ultra-endurance events are becoming increasing popular. Participation in the multi-day events adds a lot of physical and mental strain on the body, while the athletes are still required to perform. Without appropriate recovery the athletes are at increased risk of overreaching, injury, or illness.

Therefore, the purpose of the study is to create a better understanding of the exercise fatigue experienced during ultra-endurance performance and the role intermittent exogenous ketosis (IEK) plays in reducing the amount of fatigue to maintain performance during multi-day racing and lower the risk of injury and illness.

Participants will first compete in a 8-day simulated stage race performed on taxc trainers and then we will conduct a field study during the Absa Cape Epic a 8-day mountain bike stage race. Immediately following each stage and 30-mins before bed the participants will consume either a ketone ester and taste-match placebo drink. During the race the following variables will be measured; hydration status, weight change, activity readiness, and nutrition intake. Cognitive function will be assessed on day 2, 4 and 8 of racing. One day before and one day after the race the participants will report to the lab to assess basal metabolic rate, stress via questionnaires, appetite, cognitive function, muscle biopsies, venous blood samples, mechanical efficiency and 30-min Time Trial.

ELIGIBILITY:
Inclusion Criteria:

* have been cycling consistently for at least 1 year before entry into the study
* have been cycling for a minimum of 7 hours per week for the 6 months leading up to the study
* additional for the field study: valid entry to the 2025 edition of the Absa Cape Epic
* non-smoker

Exclusion Criteria:

* Do not follow a ketogenic diet or low-carbohydrate diet
* Have any metabolic or auto-immune disease that will influence their metabolism
* Take medication or supplements that is known to affect ketone supplement metabolism
* suffering from a recurring injury or illness from which they have not fully recovered that is a contr-indication to perform high-intensity exercise
* Unable to finish each stage
* Women: if they are pregnant or breastfeeding

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Muscle soreness | During the intervention
  Visual analog scale (0-10) How sore does you leg muscles feel? The VAS was used as a subjective measure of muscle soreness
Physical stress | pre-intervention and 1 day after the intervention
  RESTQ-76 sport questionnaire was used to assess the stress-recovery balance
Hydration status | Baseline, During the intervention and 1 day after the intervention
  Before every stage, the participants provided a urine sample in a cup. A urine-specific refractometer (Atago) was used to determine their hydration status
Cognitive function: reaction time | Pre-intervention, day 2, 4 and 8 of the intervention
  CANTAB test battery reaction time test was used to determine reaction time in milliseconds.
Cognitive function: rapid visual processing | Pre-intervention, day 2, 4 and 8 of the intervention
  CANTAB test battery rapid visual processing test was used to assess their susceptibility to false alarms
Cognitive function: swm | Pre-intervention, day 2, 4 and 8 of the intervention
  CANTAB spatial working memory test was used to access executive function; the main outcome measure used was the number of errors
Sleep Duration | 1 week prior to racing and during the race
  Fitbit inspire 3 was used to measure sleep duration (hours:minutes:seconds)
Sleep: REM | 1 week prior to racing and during the race
  The Fitbit Inspire 3 was used to measure the total duration of rapid eye motion (REM)sleep during each night for the duration of the study. The REM sleep phase will be analysed in minutes
Sleep: Non-REM | 1 week prior to racing and during the race
  The Fitbit Inspire 3 will be used to determine the NON-REM sleep phase for each night in minutes
Sleep: WASO | 1 week prior to racing and during the race
  The FITBIT inspire 3 will be used to measure wake after sleep onset in minutes for each night

SECONDARY OUTCOMES:
Mechanical efficiency | pre-intervention and 1 day after the intervention
  Mechanical efficiency will be determined during three constant load (100 watts, 150 watts, and 200 watts) cycling bouts of 5 minutes on a calibrated ergometer (Avantronic Cyclus II). Throughout the test, gas exchange will continuously be measured using calibrated metabolic analyzer with a face mask (Cortex, Metalyzer IIIb). VO2 and VCO2 data of the final minute of each workload will be used to calculate gross efficiency (%).
Time trial performance | pre-intervention and 1 day after the intervention
  The participants will perform a 30-minute time trial. The average power output (watts) achieved will be used as the outcome measure.
Appetite | pre-intervention, during the intervention, 1 day after the intervention
  Appetite will be assessed with a Likert visual analog scale (0-10) using the following four questions:
  "How hungry do you feel?" "How full do you feel?" "How satisfied do you feel?" "How much do you think you could eat now?"
Macronutrient intake | baseline, during the intervention
  Participants will complete a food diary using the Mijnetemeter application on their phone. Total fat, protein and carbohydrate intake will be determined in grams for each day.
Total energy intake | baseline, during the intervention
  Participants will complete a food diary, using the Mijnetemeter application on their phones. total energy intake (kilojoules) will be calculated for each day.
Racing intensity | during each stage
  hear rate zones during racing
Body weight change | During the intervention
  Body mass was measured using a SECA, model 813 electrical scale, before and after each stage as a secondary method to assess hydration status. Body mass was measured to the nearest 0.1 kilogram

CONTACTS AND LOCATIONS:
Overall Officials: Chiel Poffé, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium